CLINICAL TRIAL: NCT03199755
Title: Efficacy of Dried Leaf Artemisia (DLA) Versus Coartem (ACT): A Randomized Controlled Clinical Trial for Comparing DLA vs. ACT to Treat Malaria
Brief Title: Dried Leaf Artemisia (DLA) Compared to Artemisinin Combination Therapy (ACT) vs Malaria
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn in 2018 because clinicians did not follow protocols, issues with communication and also with tablet processing, nearby Ebola outbreak in 2018 (in the N Kivu area) confounded efforts.
Sponsor: Worcester Polytechnic Institute (Other)
Collaborators: Plesion International, Coatesville, PA (Unknown); HEAL Africa Hospital, Goma, Democratic Republic of Congo (Unknown); Rwanguba Reference Hospital, Rwanguba, Democratic Republic of Congo (Unknown)
Responsible Party: Principal Investigator, Pamela Weathers, Professor of Biology and Biotechnology, Worcester Polytechnic Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-297
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Malaria
Keywords: therapeutic; ACT; gametocyte
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT (Active Comparator): Standard Artemisinin Combination Therapy (ACT) being used as currently approved antimalarial therapy at WHO and manufacturer recommended dosage. The specific ACT used is artemether-lumefantrine (Coartem). Form is scored tablets that each contain 20 mg artemether and 120 mg lumefantrine.
  Tablets per dose, are given BID for 3 days as shown below:
  Coartem tablets/dose by bodyweight; tablets/day morning and evening for total of 6 doses over 3 days
  Body weight (kg) and Tablets: 5 to <15 kg, 1 tab; 15 to <25 kg, 2 tabs; 25 to <35 kg, 3 tabs; 35 kg and over, 4 tabs.
  Interventions: Drug: ACT
- DLA1 (Experimental): Dried leaf Artemisia annua (DLA) from 0.25-1 g total/day, BID. DLA is given as 500 mg tablets according to body weight (see below) for 5 days.
  DLA tablets/dose by bodyweight; tablets/day, morning and evening, for total of 10 doses over 5 days.
  Body weight (kg) and tablets/dose:
  For DLA1x: 5 to < 15 kg, 1/4 tab; 15-30 kg, 1/2 tab; 1/2>30 kg, 1 tab.
  Interventions: Drug: DLA1
- DLA2 (Experimental): Dried leaf Artemisia annua (DLA) from 0.5-2 g total/day, BID. DLA is given as 500 mg tablets according to body weight (see below) for 5 days.
  DLA tablets/dose by bodyweight; tablets/day, morning and evening, for total of 10 doses over 5 days.
  Body weight (kg) and tablets/dose:
  For DLA2x: 5 to < 15 kg, 1/2 tab; 15-30 kg, 1 tab; >30 kg, 2 tabs.
  Interventions: Drug: DLA2

INTERVENTIONS:
Drug: ACT — Current approved drug for treating malaria
  Other Names: Coartem; artemether and lumefantrine
  Arms: ACT
Drug: DLA1 — Experimental drug treatment, single dose.
  Other Names: dried leaf artemisia
  Arms: DLA1
Drug: DLA2 — Experimental drug treatment, doubled the dose of DLA1.
  Other Names: dried leaf artemisia
  Arms: DLA2

SUMMARY:
The overall goal is to validate efficacy and potential superiority of dried leaf Artemisia annua (DLA) vs. artemisinin combination therapy (ACT) to cure malaria and to demonstrate elimination of the transmission stage (gametocytes) of the disease. This is a 3 arm trial in Democratic Republic of Congo covering 600 total adult and pediatric patients. Final validation of infection from dried blood samples will be done at WPI.

DETAILED DESCRIPTION:
A clinical trial in DR Congo to validate that oral consumption of dried leaf tablets of the plant Artemisia annua can cure malaria and prevent its transmission.

PI: Pamela Weathers, Ph.D. & Prof. of Biology and Biotechnology, Lead Institution: Worcester Polytechnic Institute, 100 Institute Rd, Worcester, MA 01609

Background:

The plant Artemisia annua produces artemisinin, which is currently extracted and purified from the plant and used to produce the current standard of antimalarial care, artemisinin combination therapy (ACT). While some human trials have been done using dried leaf Artemisia (DLA) to treat malaria, none has been extensive enough to provide evidence convincing to the key regulatory bodies, e.g. WHO. There is animal and human evidence suggesting that DLA not only is highly efficacious at low doses, but also treats ACT-resistant malaria and may inhibit development of the gametocytes, which is the blood parasite stage that enables retransmission to the next mosquito host. ACTs have not shown full efficacy in quelling transmission. Furthermore, ACT drug resistance is now confirmed in Southeast Asia and may be emerging in Africa. Thus, this study is unique, timely and needed because:

* DLA has not been studied yet in a larger human trial.
* DLA has not been compared in a human trial to the current ACT antimalarial therapy.
* DLA shows promise at inhibiting the gametocyte transmission stage of malaria and would thereby break the cycle of malaria.
* Investigators have a full supply chain in place to grow, produce and package DLA tablets in a GMP facility and have distribution channels ready to deliver the drug to pharmacies in Eastern Africa.
* Investigators' therapeutic approach is less costly than ACT and is under the control of Africans; therapeutics by and for Africans.

Specific Aims:

Investigators overall goal is to validate efficacy and potential superiority of DLA vs. ACT to cure malaria and to demonstrate elimination of the transmission stage of the disease (gametocytes). The trial has 3 specific aims:

1. Compare overall clinical outcomes efficacy of two different doses of DLA vs. standard ACT treatment.
2. Compare parasite level via Rapid Diagnostic Test (RDT) at D0 and then via microscopy at D0-D5, D14, D28 on all patients from each arm of the trial (DLA1x, DLA2x vs. ACT).
3. Compare level of gametocytes via qPCR of dried blood spots at D0, D14, D28 on a randomly selected subset of patients from each arm of trial (DLA1x, DLA2x vs. ACT).

Dried leaves of A. annua will be provided by Botanical Extracts EPZ (BEEPZ), which is a processing facility based in the Export Processing Zone (EPZ) in Athi River, Kenya. BEEPZ extracts and purifies raw material from an agricultural supply chain of A. annua grown in Kenya, Uganda, and Tanzania. The pulverized dried leaves will then be exported to Rene Industries LTD, in Kampala, Uganda. Rene is a GMP pharmaceutical facility that investigators have inspected and that will manufacture and blister pack A. annua tablets for export to DR Congo where patients at the Rwanguba Reference Hospital (North Kivu area) will be treated.

Patients in the Coartem Arm will receive the control ACT drug using the prescribed dosing regimen according to RD Congo National Protocol and by the manufacturer (TABLE 1). A single Coartem tablet contains 20 mg artemether and 120 mg lumefantrine. All ACTs will be purchased from an EU source to obviate any counterfeit ACT drugs, which can be problematic throughout Africa. Coartem is orally administered twice daily, morning and evening, for 3 days per WHO and manufacturer guidelines.

Patients in the two DLA Arms will receive the drug using the following dosing scheme (TABLE 2) based on prior successful treatment of both adults and pediatric patients with the 1x dose. A single tablet contains 500 mg A. annua DLA. Artemisinin delivered via DLA is > 40 fold more bioavailable than artemisinin delivered as pure drug, i.e. Coartem. Two doses of DLA/day are orally delivered, morning and evening, to each patient for 5 days.

TABLE 1. Coartem dosing. Coartem tablets/dose by bodyweight; tablets/day morning and evening for total of 6 doses over 3 days

Body weight (kg) and Tablets: 5 to <15 kg, 1 tab; 15 to <25 kg, 2 tabs; 25 to <35 kg, 3 tabs; 35 kg and over, 4 tabs.

TABLE 2. DLA dosing. DLA tablets/dose by bodyweight; tablets/day, morning and evening, for total of 10 doses over 5 days.

Body weight (kg) and tablets/dose:

For DLA1x: 5 to < 15 kg, 1/4 tab; 15-30 kg, 1/2 tab; 1/2>30 kg, 1 tab. For DLA2x: 5 to < 15 kg, 1/2 tab; 15-30 kg, 1 tab; >30 kg, 2 tabs.

Duration:

The 600 human subjects will be recruited over 2-3 months in DRC where participants will be treated. Dried blood samples collected over the duration of the study will be sent to WPI where the Weathers lab will extract parasite RNA and analyze via qPCR for gametocytes. The entire trial and PCR analyses are anticipated to take no more than 18 months.

Plesion International a Pennsylvania NGO has long term contacts with Prof. Weathers at WPI, the DRC hospital, DRC doctors, the Ugandan GMP manufacturing facility, and now also with BEEPZ. Plesion will manage all aspects of the African interactions and subcontract to WPI who will manage the overall project under Prof. Weathers direction.

ELIGIBILITY:
Inclusion Criteria:

* Positive RDT for malaria and
* Positive blood smear for malaria.

Exclusion Criteria:

* All pregnant mothers less than 12 weeks gestational age.
* Children weighing less than 5 kg.
* Patients who have taken any antimalarial immediately prior to study admission.
* All patients with any form of severe malaria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in gametocyte reduction/elimination | Day 28 for both microscopic and qPCR measurements.
  Use microscopy and qPCR to compare change in gametocyte carriage among the 3 treatment arms.
Change in parasitemia elimination | Day 28 for each patient.
  Use microscopy to measure and compare parasitemia elimination in the blood of patients among the 3 treatment arms.

SECONDARY OUTCOMES:
Reduced side effects by DLA vs. ACT among the 3 arms | Through 28 days for each patient.
  Compare patient side effects observationally measured among the 3 treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Weathers, PhD, Principal Investigator — WPI
Locations (1):
- Rwanguba Reference Hospital, Goma, North Kivu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided